CLINICAL TRIAL: NCT04106362
Title: Randomized Phase II Trial of Radiotherapy With Concurrent Cisplatin +/- Concurrent Cetuximab for HPV-Positive Oropharyngeal Squamous Cell Carcinoma (OPSCC) in KRAS-Variant Patients
Brief Title: Radiation Therapy and Cisplatin With or Without Cetuximab in Treating Patients With HPV Positive, KRAS-Variant Stage III-IV Oropharyngeal Squamous Cell Carcinoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: low enrollment
Sponsor: Jonsson Comprehensive Cancer Center (Other)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 19-000543; NCI-2019-03636 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2019-09-25; First posted 2019-09-27 (Actual); Last update posted 2023-06-01 (Actual); Status verified 2023-05

CONDITIONS: Clinical Stage III HPV-Mediated (p16-Positive) Oropharyngeal Carcinoma AJCC v8; Clinical Stage IV HPV-Mediated (p16-Positive) Oropharyngeal Carcinoma AJCC v8; KRAS Protein Variant; Pathologic Stage III HPV-Mediated (p16-Positive) Oropharyngeal Carcinoma AJCC v8; Pathologic Stage IV HPV-Mediated (p16-Positive) Oropharyngeal Carcinoma AJCC v8
MeSH Terms: conditions — Oropharyngeal Neoplasms | interventions — Cetuximab; Cisplatin; 1,2-diaminocyclohexaneplatinum II citrate; Platinum; Radiotherapy; Radiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Arm I (radiation therapy, cisplatin) (Active Comparator): Beginning on day 0, patients undergo radiation therapy over 6 weeks for a total of 35 fractions. Patients also receive cisplatin IV over 1-2 hours on days 0 and 21.
  Interventions: Drug: Cisplatin; Other: Quality-of-Life Assessment; Other: Questionnaire Administration; Radiation: Radiation Therapy
- Arm II (cetuximab, radiation therapy, cisplatin) (Experimental): Patients receive cetuximab IV over 120 minutes 5-7 days prior to start of radiation therapy and then IV over 60 minutes weekly on Monday or Tuesday for 7 weeks. Patients also undergo radiation therapy and receive cisplatin as in Arm I.
  Interventions: Biological: Cetuximab; Drug: Cisplatin; Other: Quality-of-Life Assessment; Other: Questionnaire Administration; Radiation: Radiation Therapy

INTERVENTIONS:
Biological: Cetuximab — Given IV
  Other Names: Cetuximab Biosimilar CDP-1; Cetuximab Biosimilar CMAB009; Cetuximab Biosimilar KL 140; Chimeric Anti-EGFR Monoclonal Antibody; Chimeric MoAb C225; Chimeric Monoclonal Antibody C225; Erbitux; IMC-C225
  Arms: Arm II (cetuximab, radiation therapy, cisplatin)
Drug: Cisplatin — Given IV
  Other Names: Abiplatin; Blastolem; Briplatin; CDDP; Cis-diammine-dichloroplatinum; Cis-diamminedichloridoplatinum; Cis-diamminedichloro Platinum (II); Cis-diamminedichloroplatinum; Cis-dichloroammine Platinum (II); Cis-platinous Diamine Dichloride; Cis-platinum; Cis-platinum II; Cis-platinum II Diamine Dichloride; Cismaplat; Cisplatina; Cisplatinum; Cisplatyl; Citoplatino; Citosin; Cysplatyna; DDP; Lederplatin; Metaplatin; Neoplatin; Peyrone''s Chloride; Peyrone''s Salt; Placis; Plastistil; Platamine; Platiblastin; Platiblastin-S; Platinex; Platinol; Platinol- AQ; Platinol-AQ; Platinol-AQ VHA Plus; Platinoxan; Platinum; Platinum Diamminodichloride; Platiran; Platistin; Platosin
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Ancillary studies
Radiation: Radiation Therapy — Undergo radiation therapy
  Other Names: Cancer Radiotherapy; Irradiate; Irradiated; irradiation; Radiation; Radiotherapeutics; RADIOTHERAPY; RT; Therapy, Radiation

SUMMARY:
This phase II trial studies how well radiation therapy and cisplatin with or without cetuximab works in treating patients with human papillomavirus (HPV) positive, KRAS-variant stage III-IV oropharyngeal squamous cell carcinoma. Radiation therapy uses high energy x-rays to kill tumor cells and shrink tumors. Drugs used in chemotherapy, such as cisplatin, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Immunotherapy with monoclonal antibodies, such as cetuximab, may help the body?s immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread. Giving radiation therapy, cisplatin, and cetuximab may work better in treating patients with HPV positive, KRAS-variant oropharyngeal squamous cell carcinoma compared to radiation therapy and cisplatin alone.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the efficacy of radiation therapy with concurrent cisplatin combined with concurrent cetuximab in KRAS-variant oropharyngeal squamous cell carcinoma (OPSCC) patients in terms of overall survival (OS) at 2 years.

SECONDARY OBJECTIVES:

I. To determine the efficacy of radiation therapy with concurrent cisplatin combined with concurrent cetuximab in KRAS-variant OPSCC patients in terms of patterns of failure at 6 months and 2 years.

II. To determine the efficacy of radiation therapy with concurrent cisplatin combined with concurrent cetuximab in KRAS-variant OPSCC patients in terms of progression-free survival (PFS) at 2 years.

III. To determine the efficacy of radiation therapy with concurrent cisplatin combined with concurrent cetuximab in KRAS-variant OPSCC patients in terms of locoregional control (LRC) at 2 years.

IV. To determine the efficacy of radiation therapy with concurrent cisplatin combined with concurrent cetuximab in KRAS-variant OPSCC patients in terms of distant metastasis-free survival (DMFS) at 2 and 5 years.

V. To determine the efficacy of radiation therapy with concurrent cisplatin combined with concurrent cetuximab in KRAS-variant OPSCC patients in terms of OS at 5 years.

VI. To determine the safety of radiation therapy with concurrent cisplatin combined with concurrent cetuximab in KRAS-variant OPSCC patients in terms of acute toxicity profiles at the end of radiation, at 1 month, and at 6 months.

VII. To determine the safety of radiation therapy with concurrent cisplatin combined with concurrent cetuximab in KRAS-variant OPSCC patients in terms of late toxicity profiles at 1 and 2 years.

VIII. To determine the safety of radiation therapy with concurrent cisplatin combined with concurrent cetuximab in KRAS-variant OPSCC patients in terms of patient-reported swallowing outcomes at 6 months and 1 and 2 years.

IX. To assess the predictive value of fludeoxyglucose (FDG)-positron emission tomography (PET) at 10-14 weeks post-treatment.

X. To assess the predictive value of additional blood and tissue biomarkers for disease outcomes at 2 years.

EXPLORATORY OBJECTIVES:

I. To evaluate the impact of cetuximab on the immune response as well as treatment outcome and toxicity.

II. To evaluate biomarkers for immune response in HPV-associated OPSCC through saliva and blood samples to be collected prior to treatment and at each follow-up visit.

III. To evaluate for additional checkpoint targets through tumor tissue taken at the time of initial biopsy and profiled for tumor infiltrating lymphocytes, activation markers, and antigen-specific T-cell receptor (TCR) utilization/diversity.

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM I: Beginning on day 0, patients undergo radiation therapy over 6 weeks for a total of 35 fractions. Patients also receive cisplatin intravenously (IV) over 1-2 hours on days 0 and 21.

ARM II: Patients receive cetuximab IV over 120 minutes 5-7 days prior to start of radiation therapy and then IV over 60 minutes weekly on Monday or Tuesday for 7 weeks. Patients also undergo radiation therapy and receive cisplatin as in Arm I.

After completion of study treatment, patients are followed up at 2-4 weeks, every 12 weeks for 2 years, and then every 3-12 months for up to 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent obtained from the patient/legal representative prior to performing any protocol-related procedures, including screening evaluation
* Newly diagnosed, untreated, biopsy-proven HPV+ squamous cell carcinoma of the oropharynx. Cytologic diagnosis from a cervical lymph node is sufficient in the presence of clinical evidence of a primary tumor in the oropharynx. Clinical evidence should be documented, may consist of palpation, imaging, or endoscopic evaluation and should be sufficient to estimate the size of the primary (for T stage). HPV-positivity will be defined as tumors that are p16-positive by immunohistochemistry
* Selective stage III-IV disease (T3-T4 or N2-N3 disease) by American Joint Committee on Cancer (AJCC) 8th edition as determined by a computed tomography (CT) scan or magnetic resonance imaging (MRI) of the head and neck, CT neck, chest, abdomen, pelvis or a PET =< 6 weeks of registration
* Confirmation of KRAS-variant status as assessed by genotyping from a cheek swab sample at MiraDx
* Lifetime cumulative smoking history of < 10 pack-years. The cumulative total of the number of pack-years during each period of active smoking is the lifetime cumulative history

  * Note: Investigators are discouraged from enrolling patients with a history of very sustained use (such as several years or more) of non-cigarette tobacco products alone given that the effect of non-cigarette tobacco products on the survival of patients with p16-positive oropharyngeal cancers is undefined
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 ? 1 within 60 days prior to registration
* Hemoglobin >= 9 g/dL (5.58 mmol/L) (within 2 weeks prior to registration)
* Absolute neutrophil count (ANC) >= 1500/uL (cells/mm^3) (within 2 weeks prior to registration)
* Platelet count >= 100,000/uL (cells/mm^3) (within 2 weeks prior to registration)
* Total bilirubin =< 1.5 mg/dL (25.65 umol/L) or =< 3.0 mg/dL if the patient has a history of Gilbert?s disease (within 2 weeks prior to registration)
* Aspartate transaminase (AST)/alanine transaminase (ALT) =< 2 x the institutional upper limit of normal (ULN) (within 2 weeks prior to registration)
* Serum creatinine =< 1.5 x institutional ULN OR creatinine clearance (measured via 24-hour urine collection) >= 50 ml/min (that is, if serum creatinine is > 1.5 times the ULN, a 24-hour urine collection to calculate creatinine clearance must be performed) (within 2 weeks prior to registration)
* Female subjects must either be of non-reproductive potential (i.e., post-menopausal by history: >= 60 years old and no menses for at least 1 year without an alternative medical cause, OR history of hysterectomy, OR history of bilateral tubal ligation, OR history of bilateral oophorectomy) or must have a negative serum pregnancy test within 7 days prior to enrollment
* Female subjects of child bearing potential and male subjects with partners of child bearing potential must agree to adequate contraceptive measures (hormonal or barrier methods) during treatment and for 2 months after the last dose of cetuximab
* Subject is willing and able to comply with the protocol for the duration of the study including undergoing treatment, scheduled visits, and examinations including follow up

Exclusion Criteria:

* Patients with biopsy-proven metastatic, HPV-negative, KRAS-variant negative, or recurrent head and neck squamous cell carcinoma (HNSCC)
* Patients with primary site of tumor outside of the oropharynx, specifically of the oral cavity, salivary glands, nasal cavity, paranasal sinuses, larynx, hypopharynx, or nasopharynx
* Patients with prior radiation therapy (RT) that would result in overlap of radiation therapy treatment fields (superficial x-ray of skin lesions excluded)
* Gross total excision (ex. tonsillectomy) of the primary tumor; however, partial removal of the tumor to alleviate an impending airway obstruction does not make the patient ineligible. Initial surgical treatment, excluding diagnostic biopsy of the primary site or nodal sampling of neck disease, as well as radical or modified neck dissection is not permitted
* Prior systemic chemotherapy or biologic therapy for the study cancer; note that prior chemotherapy or biologic therapy for a different cancer is allowable
* Prior therapy that specifically and directly targets the EGFR pathway
* History of another primary invasive malignancy except for:

  * Malignancy treated with curative intent and with no known active disease >= 3 years before the first dose of study drug and of low potential risk for recurrence
  * Adequately treated non-melanoma skin cancer or lentigo maligna without evidence of disease
  * Adequately treated low risk prostate cancer without evidence of disease
  * Adequately treated carcinoma in situ without evidence of disease e.g., cervical cancer in situ, and ductal breast carcinoma in situ (DCIS)
* History of infusion reaction or hypersensitivity to cetuximab OR allergic reactions attributed to compounds of chemical or biologic composition similar to those of cetuximab
* Documented uncontrolled intercurrent illness or co-morbidity including, but not limited to, ongoing or active bacterial or fungal infection requiring intravenous antibiotics, uncontrolled congestive heart failure, cardiomyopathy, uncontrolled hypertension, unstable angina pectoris, cardiac arrhythmia, acquired immune deficiency syndrome (AIDS) based upon current Centers for Disease Control and Prevention (CDC) definition, or psychiatric illness/social situations that would limit compliance with study requirements or compromise the ability of the subject to give written informed consent
* Female subjects who are pregnant or breastfeeding as well as male or female patients of reproductive potential who are not employing an effective method of birth control
* Patients with clinically relevant coronary artery disease or history of myocardial infarction in the last 12 months or high-risk of uncontrolled arrhythmia or uncontrolled cardiac insufficiency
* Patients with uncontrolled or poorly-controlled hypertension (> 180 mmHg systolic or > 130 mmHg diastolic)
* Any condition that, in the opinion of the investigator, would interfere with evaluation of study treatment or interpretation of patient safety or study results
* Involvement in the planning and/or conduct of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2020-01-14 (Actual); Primary Completion 2023-05-23 (Actual); Study Completion 2023-05-23 (Actual)

PRIMARY OUTCOMES:
Overall survival (OS) | From time of randomization to death due to any cause, assessed at 2 years
  OS will be estimated in each study arm by Kaplan-Meier estimate. Summaries of the number and percentage of patients who have died, are still in survival follow-up, are lost to follow-up and have withdrawn consent will be provided along with median OS. Furthermore, a binomial test of proportions will be used to test difference in 2-year OS between the two arms. Exact tests and continuity correction strategies will be considered when appropriate.

SECONDARY OUTCOMES:
Primary tumor control | Up to 5 years
  Will be determined by Response Evaluation Criteria in Solid Tumors version (v). 1.1. Kaplan-Meier estimate will be used to describe primary control rate for each arm. Furthermore, log-rank test will be used to test the difference between primary tumor control between the two arms.
Locoregional recurrence rate | Up to 5 years
  Will be determined by surveillance imaging, with failure defined as appearance of new disease in the head and neck from the date of randomization. Kaplan-Meier estimate will be used to describe locoregional recurrence rate for each arm. Furthermore, log-rank test will be used to test difference in locoregional recurrence rates between the two arms.
Acute toxicity | Up to 5 years
  Will be evaluated using the Common Terminology Criteria for Adverse Events (CTCAE) v5.0. The safety analysis set will be used for safety analyses. The overall safety and tolerability will be assessed throughout the study period. All adverse event (AE) data will be listed individually by treatment group and patient identifier.
Late toxicity | Up to 5 years
  Will be evaluated using the CTCAE v5.0. The safety analysis set will be used for safety analyses. The overall safety and tolerability will be assessed throughout the study period. All AE data will be listed individually by treatment group and patient identifier.

OTHER OUTCOMES:
Germline mutation prediction rate | Up to 5 years
  Will assess if additional germline mutations predict rate of progression free survival (PFS), overall survival and toxicity. Multivariate Cox proportional hazards models will be used to assess if the endpoint is a prognostic variable for PFS, OS after adjusting for treatment arms and other clinical variables. Multivariate logistic regression model will be used to evaluate the association with toxicity.
Nonsynonymous mutational load and intratumoral heterogeneity clinical outcome predictions | Up to 5 years
  Will assess if nonsynonymous mutational load and intratumoral heterogeneity are predictive markers for clinical outcome (progression-free survival, overall survival, and toxicity) using next generation sequencing of baseline and relapsed tumors. Multivariate Cox proportional hazards models will be used to assess if the endpoint is a prognostic variable for PFS, OS after adjusting for treatment arms and other clinical variables. Multivariate logistic regression model will be used to evaluate the association with toxicity.
Change in circulating lymphocytes | Baseline up to 5 years
  Will assess changes to circulating lymphocytes including CD-8, T-regulatory cells, and myeloid suppressor cells before, during and after treatment and correlations with progression free-survival, overall survival and toxicity. Multivariate Cox proportional hazards models will be used to assess if the endpoint is a prognostic variable for PFS, OS after adjusting for treatment arms and other clinical variables. Multivariate logistic regression model will be used to evaluate the association with toxicity.

CONTACTS AND LOCATIONS:
Overall Officials: Robert K Chin, Principal Investigator — UCLA / Jonsson Comprehensive Cancer Center
Locations (1):
- UCLA / Jonsson Comprehensive Cancer Center, Los Angeles, California, United States